CLINICAL TRIAL: NCT00898924
Title: Evaluation of EGFR and K-ras Mutations in Patients With Stage III NSCLC Treated on CALGB 30106
Brief Title: Epidermal Growth Factor Receptor and K-ras Mutations in Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150508; U10CA031946 (NIH); CALGB-150508; CDR0000491128 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Molecular Diagnostic Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue, whole blood and serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Tissue samples were collected from patients on Day 1, Cycle 1. Whole blood and serum samples were collected on Day 1 (Cycle 1), Day 1 (Cycle 3), post-radiotherapy ZD1839 and at progression.
  Interventions: Genetic: molecular diagnostic method; Genetic: mutation analysis

INTERVENTIONS:
Genetic: molecular diagnostic method
Genetic: mutation analysis

SUMMARY:
RATIONALE: Collecting and storing samples of tissue from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at epidermal growth factor receptor mutations and k-ras oncogene mutations in patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of epidermal growth factor receptor (EGFR) and K-ras mutations in patients with stage III non-small cell lung cancer (NSCLC) treated on CALGB 30106.
* Correlate presence or absence of EGFR and/or K-ras mutations with radiographic response to treatment in these patients.

OUTLINE: Tissue samples are analyzed for epidermal growth factor receptor and K-ras mutations.

ELIGIBILITY:
Inclusion criteria:

1. Eligible patients had histologic documentation of un- treated stage III NSCLC.
2. Radiation oncologist confirmation was required that radiation could be given per protocol.
3. Eastern Cooperative Group Criteria Performance Status of 0 to 2
4. Tumor specimen paraffin block or unstained slides and standard initial laboratory tests
5. Signed institutional review board-approved, protocol-specific in- formed consent in accordance with federal and institutional guidelines

Exclusion criteria:

1. Patients with scalene, supraclavicular, or contralateral hilar lymph node involvement, or direct invasion of the vertebral body or with a pleural effusion were ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stage III non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2006-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 3 years
Progression free survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pasi Janne, MD, PhD, Study Chair — Dana-Farber Cancer Institute